CLINICAL TRIAL: NCT06207058
Title: Evaluation of a Screen and Treat Protocol for Influenza in Socially Vulnerable Communities.
Brief Title: Evaluation of a Screen and Treat Protocol for Influenza
Status: Terminated | Type: Observational
Why Stopped: Limited enrollment opportunities due to low rates of viral infections
Sponsor: Tricore, Inc (Other)
Responsible Party: Sponsor
Other Study IDs: Tricore
Record Dates: First submitted 2024-01-05; First posted 2024-01-16 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Influenza Positive: Subjects testing positive will receive baloxavir marboxil as a single oral dose as soon as possible and within 48-hours of influenza symptom onset. Dosing will be delivered based on the package insert
  Interventions: Drug: Baloxavir Marboxil
- Influenza Negative: Subjects testing negative for influenza will have no drug administered

INTERVENTIONS:
Drug: Baloxavir Marboxil — Subjects testing positive for influenza will receive a dose of Baloxavir Marboxil orally, according to the dosing indicated in the package insert.
  Groups: Influenza Positive

SUMMARY:
This study seeks to demonstrate that the laboratory can mitigate respiratory virus transmission in underserved populations by using laboratory data to identify communities at risk for increase vial activity (hot spots) and intervening with a test-to-treat model provides increased access to influenza diagnostics and treatment in vulnerable and underserved communities.

DETAILED DESCRIPTION:
The investigators have developed an analytic algorithm that uses measures from the CDC COVID-19 Hot Spot Criteria and Brown University School of Public Health to determine COVID-19 and Influenza Hot Spots and Testing Deserts, respectively. The Hot Spot designation was based on the CDC county-specific Hot Spot criteria that has been used to deploy resources for interventions (i.e., laboratory testing, community mitigation, health communications and health care) specific needs for the communities of interest. The CDC hot spot criteria is based on COVID-19 rates at the county level. The adaptations to the criteria allows interventions to focus on a concentrated community and deliver the interventions in places that the community is already engaging, such as community centers, senior centers and parks.

Through collaboration with local community centers, the investigators are able to deploy a mobile testing unit to a community center, park or senior center that is in close proximity to the identified neighborhood for rapid onsite testing for Influenza A&B and SARS-CoV2 using the cobas Liat system.

New Mexico has adopted "New Mexico Board of Pharmacy Protocol for Pharmacists Prescribing of Dangerous Drugs in Conjunction with Point of Care Testing" (NMBOP POCT Protocol, Appendix 5) that allows pharmacists the prescriptive authority to prescribe Influenza antiviral therapy in conjunction with a positive point of care test (POCT). TriCore employs two (2) on-site clinical pharmacists who will follow all of the pharmacist mandates included in the regulation to prescribe and distribute Xofluza according to the approved protocol in the test-to-treat model presented in this study. The NMBOP PCOT Protocol documents the eligibility and requirements of the certified prescribing pharmacists (pharmacist) following this protocol.

The pharmacist will perform a screening physical assessment, health assessment and medical history for the patient. If the subject meets the inclusion criteria, they will have a point of care test performed. If the subject meets the exclusion criteria, they will be excluded from the study. Testing will be performed using the cobas® SARS-CoV-2 & Influenza A/B assay on the cobas® Liat® system from a self-collected nasal swab. Subjects who test positive for influenza A or B will be prescribed Xofluza with no additional refills. The pharmacist will follow-up with the patient 24-48 hours following administration for evaluation of signs/symptoms and will refer the patient to their primary care provider, provider, or clinic for recommended laboratory testing and follow-up if appropriate.

All subjects eligible for Xofluza will receive patient education and counseling on drug information, adherence, side effects, and other patient educational materials, as appropriate. All subjects eligible for influenza antiviral therapy, but having contraindications to the therapy, or do not wish to use the therapy will be referred to their primary care provider, provider, or clinic for further evaluation.

Subjects testing positive for SARS-CoV-2 will be referred by the pharmacist to the subjects' primary care provider, provider, or clinic for further medical assessment and follow-up, if appropriate. Subjects testing negative for all targets (SARS-CoV-2 and Influenza A&B) with a high index of suspicion for influenza, will be referred by the pharmacist to the subjects' primary care provider, provider, or clinic for further medical assessment and follow-up, if appropriate. All subjects will receive a follow-up call 14-days following the study visit to assess their symptom resolution and the impact of their illness on their well-being

The mobile testing unit will be deployed a minimum of 2 times per week following the determination of the influenza season by the New Mexico Department of Health. The investigators expect to screen 50-100 patients per week for the duration of the influenza season (approximately 12 weeks) for a total of 600-1,2000 patients. With an anticipated 10% positivity rate for influenza, the investigators expect at least 5-10 patients per week to be eligible for treatment for a total of 60-120 subjects eligible over the course of the study. All subjects will be provided a survey to evaluated their ability to access respiratory virus testing and their acceptance of and trust in using a mobile unit for access to treatment and therapeutics. Patients positive for SARS-CoV-2 will be counseled on options for treatment and follow up for COVID-19 infection. All subjects enrolled in the study will receive a follow-up phone call 14-days following the initial screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients: Signed informed consent by any patient capable of giving consent, or, where the patient is not capable of giving consent, by his or her legal/authorized representative.
* Adolescent patients not able to legally consent: written informed consent for study participation is obtained from patient's parents or legal guardian, with assent as appropriate by the patient, depending on the patient's level of understanding and capability to provide assent
* Age ³ 5 years at the time of signing the Informed Consent Form/Assent Form
* Ability to comply with the study protocol, in the investigator's judgment.
* Presence of (a) fever (≥38.0 °C per tympanic or rectal thermometer; ≥37.5 °C per axillary, oral or forehead/temporal thermometer) or (b) any influenza symptoms (cough, sore throat, nasal congestion, headache, feverishness or chills, muscle or joint pain, fatigue).
* The time interval between the onset of fever or influenza symptoms and the pre-dose examinations is 48 hours or less.
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse):
* Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 28 days after the last dose of study treatment. Hormonal contraceptive methods must be supplemented by a barrier method.
* A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (³ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
* Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Patients who have received more than 48 hours of antiviral treatment for the current influenza infection prior to screening
* Patients who have received Xofluza for the current influenza infection
* Known contraindication to neuraminidase inhibitors
* Patients weighing < 20 kg
* Patients unable to swallow tablets
* Patients with known severe renal impairment (estimated glomerular filtration rate < 30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis
* Patients with any of the following laboratory abnormalities detected within 24 hours prior to or during screening (according to local laboratory reference ranges:
* ALT or AST level > 5 times the upper limit of normal (ULN) or ALT or AST > 3 times the ULN and total bilirubin level > 2 times the ULN
* Pregnant or breastfeeding, or positive pregnancy test in a predose examination, or intending to become pregnant during the study or within 28 days after the last dose of study treatment
* Exposure to an investigational drug within 5 half-lives or 30 days (whichever is longer) of randomization
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Known hypersensitivity to Xofluza (baloxavir marboxil) or the drug product excipients

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals in respiratory hot spots and socially vulnerable communities identified in the algorithm.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Crossey, MD, PhD, Principal Investigator — Medical Director, Tricore Research Institute
Locations (1):
- TriCore Mobile Unit, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza Positive | Influenza Negative
Started | 1 | 24
Completed | 1 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Positive | Influenza Negative | Total
Number analyzed (Participants) | 1 | 24 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 4 | 4
  Between 18 and 65 years | 0 | 8 | 8
  >=65 years | 1 | 12 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 12
  Male | 0 | 13 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Symptom Status
Description: Patients who receive treatment are asked if symptoms are improving or worsening during the treatment follow up call, 14 days after treatment
Time Frame: 14 Days
Population: In the study timeframe, only one patient tested positive for influenza and was able to receive the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Positive | Influenza Negative
Number analyzed (Participants) | 1 | 24
Participants
  Improving | 1 | 15
  Worsening | 0 | 0
  Did not respond | 0 | 9

ADVERSE EVENTS:
Time Frame: 14 Days
Arm/Group | Influenza Positive | Influenza Negative
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/24
Other Adverse Events (participants affected / at risk) | 0/1 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT06207058/Prot_SAP_000.pdf